CLINICAL TRIAL: NCT01624311
Title: Hypothermia Treatment in Hyperammonemia and Encephalopathy
Brief Title: Pilot Study For Hypothermia Treatment In Hyperammonemic Encephalopathy In Neonates And Very Young Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uta Lichter-Konecki (Other)
Collaborators: Children's National Research Institute (Other); Medical College of Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Uta Lichter-Konecki, MD, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAN6104
Record Dates: First submitted 2012-06-13; First posted 2012-06-20 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Urea Cycle Disorders; Organic Acidemias
Keywords: High ammonia level; Hyperammonemia; Poor suck; Lethargy; Coma; Encephalopathy; Seizures; Brain edema; Urea Cycle Disorder; Ornithine Transcarbamylase Deficiency; Carbamoyl Phosphate Synthetase Deficiency; Citrullinemia; Argininosuccinic Aciduria; Organic Acidemia; Propionic Aciduria; Methylmalonic Aciduria; Isovaleric Aciduria
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Hyperammonemia; Lethargy; Coma; Brain Diseases; Seizures; Brain Edema; Ornithine Carbamoyltransferase Deficiency Disease; Carbamoyl-Phosphate Synthase I Deficiency Disease; Citrullinemia; Argininosuccinic Aciduria; Propionic Acidemia; Methylmalonic acidemia | interventions — Hypothermia, Induced; Cryotherapy; Cool-Down Exercise; Dialysis; Renal Dialysis; Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjunct Hypothermia Arm (Experimental): Patients that receive adjunct therapeutic hypothermia in addition to standard of care therapy
  Interventions: Other: Therapeutic Hypothermia
- Historic Controls (Other): Patients that were treated with standard of care therapy for the same conditions at the sponsoring institution over the past 10 years.
  Interventions: Other: Standard of Care Therapy

INTERVENTIONS:
Other: Therapeutic Hypothermia — After obtaining written consent, patients are cooled to 33.5°C (+/- 1°C ) for 72 hours and and then rewarmed by 0.5°C per every 3 hours over 18 hours.
  Other Names: Hypothermia; Hypothermia Therapy; Cooling
  Arms: Adjunct Hypothermia Arm
Other: Standard of Care Therapy — Patients with hyperammonemia and encephalopathy requiring renal replacement therapy due to a urea cycle disorder or organic acidemia that were treated at Children's National Medical Center over the past 10 years.
  Other Names: Dialysis; Hemodialysis; CVVH; CVVHD
  Arms: Historic Controls

SUMMARY:
This is a pilot study which will test the safety and feasibility of hypothermia treatment as adjunct therapy to conventional treatment of hyperammonemic encephalopathy (HAE) in neonates versus conventional treatment (dialysis, nutritional therapy, and ammonia scavenging drugs) only. The endpoint of the pilot study will be reached when either 24 patients have been enrolled and no serious adverse events were observed, when no patient has been enrolled in 5 years, or when serious adverse events occur which are clearly linked to the use of hypothermia. These would be serious complications not seen in patients on conventional therapy (dialysis , nutritional therapy, ammonia scavenging drugs) for HAE.

DETAILED DESCRIPTION:
Children with neonatal onset Urea Cycle Disorders or Organic Acidemias develop hyperammonemia (high ammonia levels) and fall into coma often causing brain damage. For these children to be able to benefit maximally from available long-term treatment and solid organ transplant, outcome of the neonatal onset crisis must be improved. Animal experiments and small clinical trials have indicated that hypothermia protects the brain during hyperammonemia. This pilot study investigates whether adjunct hypothermia therapy in addition to standard of care treatment is feasible and safe in babies with high ammonia levels in coma.

ELIGIBILITY:
Inclusion Criteria:

* Newborns >36 wks gestation and ≥2200g birth weight without co-morbidity (see exclusion criteria) that have clinical signs and symptoms of an Urea Cycle Disorders or Propionic , Methylmalonic, or Isovaleric acidemia and hyperammonemia and encephalopathy requiring renal replacement therapy.

Exclusion Criteria:

* Patients with hyperammonemia that have clinical signs and symptoms of lysinuric protein intolerance, mitochondrial disorders, congenital lactic acidosis, and fatty acid oxidation disorders, patients with rare and unrelated serious comorbidities and other genetic diseases, e.g., Down syndrome, intraventricular hemorrhage in the newborn period, traumatic brain injury, and low birth weight (<2,200 g at >36 wks gestation).
* Infants in extremis for which no additional intensive therapy will be offered by the attending neonatologist.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with unexpected Serious Adverse Events as a Measure of Safety and Tolerability | Participants will be followed for the duration of the hospital stay, an expected average of 5 weeks
  The DSMB meets within 3 weeks of each case, no later than 5 weeks after initiation of hypothermia therapy and assesses the safety and feasibility of adjunct hypothermia treatment in this patient group. The treatment of neonates and very young infants in hyperammonemic coma is very complex and adding hypothermia therapy to this treatment could not be feasible, the pilot study therefore also assesses the feasibility of adding hypothermia therapy to the standard of care treatment.
Feasibility of hypothermia therapy as adjunct therapy to the complex standard of care therapy | During the first 72h of treatment
  The standard of care therapy is very complex. It includes renal replacement therapy, metabolic diet intervention, and ammonia scavenger use. The pilot study will assess primarily for the first 72 hours of treatment and secondarily for the duration of the hospital stay, an expected average of 5 weeks, whether adding hypothermia to this already complex treatment is feasible.

SECONDARY OUTCOMES:
Time to normalization of ammonia level | During the first 72 hours of treatment
  One of the effects of hypothermia treatment is an overall slowing of metabolism which should cause less ammonia to be produced. If this is correct this should lead to a faster normalization of the ammonia level by renal replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Uta Lichter-Konecki, MD, PhD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Columbia University, Morgan Stanley Children's Hospital, New York, New York
  - Medical College Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: National Urea Cycle Disorders Foundation (Family Organisation) — http://www.nucdf.org/